CLINICAL TRIAL: NCT00114543
Title: A Randomized Trial of Aggressive or Conservative Phototherapy for Extremely Low Birth Weight Infants
Brief Title: Trial of Aggressive Versus Conservative Phototherapy in Infants <1,000 Grams Birth Weight
Acronym: Phototherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Brenda H. Morris, Lead Principal Investigator, University of Texas Health Science Center at Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NICHD-NRN-0029; M01RR016587 (NIH); M01RR000030 (NIH); M01RR000032 (NIH); M01RR000039 (NIH); M01RR000044 (NIH); M01RR006022 (NIH); M01RR000633 (NIH); M01RR000070 (NIH); M01RR007122 (NIH); M01RR000750 (NIH); M01RR000080 (NIH); M01RR008084 (NIH); U01HD036790 (NIH); U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD021397 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD040461 (NIH); U10HD040492 (NIH); U10HD040498 (NIH); U10HD040521 (NIH); U10HD040689 (NIH)
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2017-09

CONDITIONS: Hyperbilirubinemia, Neonatal; Jaundice, Neonatal; Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature
Keywords: NICHD Neonatal Research Network; Bilirubin; Phototherapy; Very Low Birth Weight (VLBW); Extremely Low Birth Weight (ELBW); Prematurity; Neurodevelopmental outcome
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aggressive ELBW (Active Comparator): In Aggressive group 1, infants with birth weights 501-750g.
  Interventions: Procedure: Aggressive Phototherapy 501-750g
- Aggressive VLBW (Active Comparator): In the Aggressive group 2, infants with birth weights 751-1000g.
  Interventions: Procedure: Aggressive Phototherapy 751-1000g
- Conservative ELBW (Active Comparator): In the Conservative group 1, infants with birth weights 501-750g.
  Interventions: Procedure: Conservative Phototherapy 501-750g
- Conservative VLBW (Active Comparator): In the Conservative group 2, infants with birth weights 751-1000g.
  Interventions: Procedure: Conservative Phototherapy 751-1000g

INTERVENTIONS:
Procedure: Aggressive Phototherapy 501-750g — Phototherapy started, stopped, and/or restarted when total serum bilirubin levels reach 5 mg/dl during days of life 1-14.
  Arms: Aggressive ELBW
Procedure: Aggressive Phototherapy 751-1000g — Phototherapy started, stopped, and/or restarted when total serum bilirubin levels reach 5 mg/dl during days of life 1-7, and started, stopped, and/or restarted when levels reach 7 mg/dl during days of life 8-14.
  Arms: Aggressive VLBW
Procedure: Conservative Phototherapy 501-750g — Phototherapy started, stopped, and/or restarted when total serum bilirubin levels reach ≥8.0 mg/dl during days of life 1-14.
  Arms: Conservative ELBW
Procedure: Conservative Phototherapy 751-1000g — Phototherapy started, stopped, and/or restarted when total serum bilirubin levels reach ≥10.0 mg/dl during days of life 1-14.
  Arms: Conservative VLBW

SUMMARY:
This multi-center, randomized clinical trial compared different bilirubin levels as thresholds for timing of phototherapy in extremely low birth weight infants. The primary hypothesis was that there would be no difference in death or neurodevelopmental impairment at 18-22 months corrected age in infants treated by either aggressive or conservative threshold limits. 1,978 infants were enrolled.

DETAILED DESCRIPTION:
In NICHD Neonatal Research Network (NRN) centers in 2002, phototherapy was administered to 94 percent of the extremely low birth weight (ELBW) infants who survive more than 12 hours. Yet, it is unclear what level of bilirubin in the blood is harmful for these very tiny infants -- no data existed from large or recent clinical trials to define the risks, benefits, and appropriate indications for phototherapy in these infants. The largest and most recent trial was the NICHD Collaborative Phototherapy Trial which involved infants treated in 1974-1976 and included only 77 ELBW infants. Data from this study and others suggested that phototherapy could have important hazards as well as benefits for ELBW infants.

This NRN study used two different bilirubin levels as thresholds for timing of phototherapy in 1,978 extremely low birth weight infants, examining the primary hypothesis that there would be no difference in death or neurodevelopmental impairment at 18-22 months corrected age between the aggressively and conservatively treated groups.

Enrolled infants were stratified by birth weight (501-750g and 751-1,000g) and randomized to receive phototherapy regimens based on either an aggressive threshold or a conservative threshold of total serum bilirubin.

In the Aggressive group:

* 501-750 grams birth weight infants, phototherapy was started, stopped, and restarted based on a total serum bilirubin threshold level of 5 mg/dl for day of life 1-14.
* 751-1,000 grams birth weight infants, phototherapy was started, stopped, and restarted based on a total serum bilirubin threshold level of 5 mg/dl for day of life 1-7 and 7 mg/dl for day of life 8-14.

In the Conservative group:

* 501-750 grams birth weight infants, phototherapy was started, stopped, and restarted based on a total serum bilirubin threshold level of 8 mg/dl for day of life 1-14.
* 751-1,000 grams birth weight infants, phototherapy was started, stopped, and restarted based on a total serum bilirubin threshold level of 10 mg/dl for day of life 1-14.

The phototherapy regimens are designed to fall within the range of clinical practice and to assure a sizable difference between groups in total serum bilirubin levels and duration of phototherapy.

The primary outcome was death or neurodevelopmental impairment at 18-22 months corrected age determined at an outpatient clinic visit. Secondary outcomes included death, abnormal neurodevelopmental outcome, severe hearing loss, cerebral palsy, blindness, and important medical outcomes.

ELIGIBILITY:
Inclusion criteria:

* 501-1000 grams birth weight
* 12-36 hours postnatal age

Exclusion criteria:

* Terminal condition (pH <6.8 for >2 hours OR persistent bradycardia, heart rate <100 bpm, associated with hypoxia for >2 hours]
* Prior use of phototherapy
* Major congenital anomaly
* Hydrops fetalis or severe hemolytic disease diagnosed in-utero
* Overt congenital nonbacterial infection
* Parental refusal or inability to provide consent
* Attending physician refusal
* Parents who are considered unlikely to return for follow-up evaluation

Ages: 12 Hours to 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1974 (Actual)
Dates: Start 2002-09; Primary Completion 2005-04 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Death or neurodevelopmental impairment (MDI <70; PDI <70; cerebral palsy; blindness; or severe hearing loss) | 0-22 months corrected age

SECONDARY OUTCOMES:
Patent ductus arteriosus requiring drug or surgical treatment | 36 weeks post conceptual age
Retinopathy of prematurity | 36 weeks post conceptual age
Bronchopulmonary dysplasia (BPD) | 36 weeks post conceptual age
Ventilator settings and FiO2 at 36 weeks | 36 weeks post conceptual age
Necrotizing enterocolitis (NEC) | 120 days old or at discharge
Intraventricular hemorrhage (IVH) by grade | 120 days old or at discharge
Periventricular leukomalacia | 120 days old or at discharge
Sepsis | 120 days old or at discharge
Hearing assessments | 120 days old or at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Ronnie Guillet, MD PhD, Principal Investigator — University of Rochester; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Barbara J. Stoll, MD, Principal Investigator — Emory University; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Brenda H. Morris, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University; Shahnaz Duara, MD, Principal Investigator — University of Miami; T. Michael O'Shea, MD MPH, Principal Investigator — Wake Forest University
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Result] Morris BH, Oh W, Tyson JE, Stevenson DK, Phelps DL, O'Shea TM, McDavid GE, Perritt RL, Van Meurs KP, Vohr BR, Grisby C, Yao Q, Pedroza C, Das A, Poole WK, Carlo WA, Duara S, Laptook AR, Salhab WA, Shankaran S, Poindexter BB, Fanaroff AA, Walsh MC, Rasmussen MR, Stoll BJ, Cotten CM, Donovan EF, Ehrenkranz RA, Guillet R, Higgins RD; NICHD Neonatal Research Network. Aggressive vs. conservative phototherapy for infants with extremely low birth weight. N Engl J Med. 2008 Oct 30;359(18):1885-96. doi: 10.1056/NEJMoa0803024. PMID 18971491
- [Result] Ahlfors CE, Vreman HJ, Wong RJ, Bender GJ, Oh W, Morris BH, Stevenson DK; Phototherapy Subcommittee; National Institute of Child Health and Development (NICHD) Neonatal Research Network. Effects of sample dilution, peroxidase concentration, and chloride ion on the measurement of unbound bilirubin in premature newborns. Clin Biochem. 2007 Feb;40(3-4):261-7. doi: 10.1016/j.clinbiochem.2006.09.006. Epub 2006 Sep 29. PMID 17069786
- [Result] Bender GJ, Cashore WJ, Oh W. Ontogeny of bilirubin-binding capacity and the effect of clinical status in premature infants born at less than 1300 grams. Pediatrics. 2007 Nov;120(5):1067-73. doi: 10.1542/peds.2006-3024. PMID 17974745
- [Result] Oh W, Stevenson DK, Tyson JE, Morris BH, Ahlfors CE, Bender GJ, Wong RJ, Perritt R, Vohr BR, Van Meurs KP, Vreman HJ, Das A, Phelps DL, O'Shea TM, Higgins RD; NICHD Neonatal Research Network Bethesda MD. Influence of clinical status on the association between plasma total and unbound bilirubin and death or adverse neurodevelopmental outcomes in extremely low birth weight infants. Acta Paediatr. 2010 May;99(5):673-678. doi: 10.1111/j.1651-2227.2010.01688.x. Epub 2010 Jan 25. PMID 20105142
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/